CLINICAL TRIAL: NCT01654354
Title: Comparison of NEOVIST 370 INJ.(Iopromide 768.86mg) With Ultravist 370 INJ.(Iopromide 768.86mg) in Abdominal CT
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Eun Cheon, Associate Professor in Radiology(Pediatric Radiology), Seoul National University Hospital
Other Study IDs: Neovist IIT
Record Dates: First submitted 2012-07-20; First posted 2012-07-31 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Abdominal CT
Keywords: Qualitative Evaluation of abdominal CT image using 4 point scale: Excellent(4)/ Good(3) / Fair(2) / Unacceptable(1)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days

INTERVENTIONS:
Drug: NEOVIST 370 INJ.(Iopromide 768.86mg)
Drug: Ultravist 370 INJ.(Iopromide 768.86mg)

SUMMARY:
Comparison of NEOVIST 370 INJ.(Iopromide 768.86mg) with Ultravist 370 INJ.(Iopromide 768.86mg) in abdominal CT

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 75 years old.
* Subjects who need CT scan
* Subjects who are willing to participate in the study and to write the informed consent form.

Exclusion Criteria:

* Subjects with severe hepatopathy whose AST or ALT ≥ 1,000 IU/L, Subjects with liver cirrhosis whose AST or ALT ≥ UNL(upper normal limit) X 3
* Severe disorder of thyroid gland
* homocystinuria
* pregnant or breastfeeding female subjects, or female subjects with childbearing potential who are not willing to use proper contraception methods
* Participation in another clinical trial within 30days of enrollment into this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who performed scheduled CT scan, mostly postoperative state of stomach cancer
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
imaging quality | end of study enrollment
  Two readers evaluate image quality of the abdomen CT by four-points scale
Adverse reaction | immediate after CT scan

SECONDARY OUTCOMES:
SNR (signal to noise ratio) / CNR (contrast to noise ratio) | at the end or enrollment
  ROI measurement at abdominal aorta and liver